CLINICAL TRIAL: NCT03184649
Title: The Effect of Ibuprofen, Paracetamol Versus Placebo on Pain During Local Anesthetic Injection and Following Dental Extraction in Primary Molars: A Randomized Clinical Trial
Brief Title: Ibuprofen, Paracetamol Versus Placebo on Pain During Local Anesthetic Injection (RCT)
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Rehab Abdelrahman Elshenawy, Principle investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: RAElshenawy
Record Dates: First submitted 2017-06-09; First posted 2017-06-12 (Actual); Last update posted 2017-06-14 (Actual); Status verified 2017-06

CONDITIONS: Analgesic Drugs; Pain Relief
MeSH Terms: interventions — Ibuprofen; Acetaminophen

STUDY DESIGN:
Intervention Model Description: three groups, two for intervention and one for comparative group
Masking Description: statistician will be blind only
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- intervention arm (Experimental): Ibuprofen suspension (Ibufen®, 100 mg/5 mL; fruit flavored, orange colour, Abbott) will be given 30 min before injection of local anesthesia. Then pain scores will be recorded from 0-4.
  Interventions: Drug: Ibuprofen
- intervention (Experimental): Paracetamol (Calpol™, 250 mg/5 mL; fruit flavored, orange color, GlaxoSmithKline) will be given 60 min before injection of local anesthesia.Then pain scores will be recorded from 0-4.
  Interventions: Drug: paracetamol
- comparator (Placebo Comparator): A fruit-flavored orange color placebo solution will be given 60 min before injection of local anesthesia.Then pain scores will be recorded from 0-4.
  Interventions: Dietary Supplement: A fruit-flavored orange color placebo solution

INTERVENTIONS:
Drug: Ibuprofen — It is a pre-analgesic will be taken before painful procedures.
  Other Names: Ibufen®
  Arms: intervention arm
Drug: paracetamol — it is a pre-analgesic drug will be taken before painful procedure.
  Other Names: calpol®
  Arms: intervention
Dietary Supplement: A fruit-flavored orange color placebo solution — orange juice as a comparative group.
  Other Names: orange juice
  Arms: comparator

SUMMARY:
The Effect of Ibuprofen, Paracetamol versus Placebo on Pain during Local Anesthetic Injection and Following Dental Extraction in Primary Molars: A Randomized clinical trial

DETAILED DESCRIPTION:
1. Diagnosis:

1. Diagnostic chart will be filled with personal, medical and dental history. DMF and def.
2. Clinical examination (intra oral and extra oral) will be done by mirror and probe to assess the inclusion criteria. All materials will be packaged in sterilizations wraps and autoclave following the required bio safety standards.

2. Intervention:

Experimental Groups:

Group 1: Ibuprofen suspension (Ibufen®, 100 mg/5 mL; fruit flavored, orange colour, Abbott). Group 2: Paracetamol (Calpol™, 250 mg/5 mL; fruit flavored, orange color, GlaxoSmithKline).

Comparative Group:

Group 3: A fruit-flavored orange color placebo solution.

Clinical procedure:

1. The drugs in all of the groups will be prepared in a fruit-flavored solution of the same color and scent.
2. Patients will be blind to one of the three pre-treatment drug groups.
3. Containers of each solution will be prepared and number-coded with the slips of paper by the assistant supervisor. The containers will be the same for all treatment groups except for the number coded with slips of paper.
4. Both the researcher and the child/parent will be blind to the content of the container.
5. The assigned solution will be taken by the patient at various times before administration of the local anesthetic agent. Ibuprofen 30 min before injection of local anesthesia paracetamol 60 min before injection of local anesthesia Placebo solution 60 min before injection of local anesthesia
6. The time of the preoperative solution administration will be recorded on the data sheet.
7. Topical anesthesia in the form of benzocaine gel 20% will be applied to the dried mucosa. All the children will be given 2% lidocaine with a 1:80,000 epinephrine injection for local anesthesia sufficient for obtaining adequate anesthesia.
8. All teeth will be extracted with a minimum of surgical trauma in an uncomplicated fashion.

Recording data

1. Pain scores will be recorded in the Pediatric Dental Clinic using a five-face scale that had been previously validated.
2. This scale has shown good construct validity as a self-report pain measure. It measures an affective dimension of a child's pain experience after injection and teeth extraction and is used in children aged 7-12 years.
3. It is easy to use and giving consistent scores from 0 to 4. It can be used for the subjective evaluation of feelings after the performance of painful dental procedures.
4. The child will be shown to a set of five cartoon faces with varying facial expressions ranging from a smile/laughter to tears. The scores given are: (0) No sign of pain. (1) Mild pain. (2) Moderate pain. (3) Severe pain. (4) Very severe pain.

ELIGIBILITY:
Inclusion Criteria:

1. Children aged 7-12 years who need extractions under local anesthesia.
2. Those having a parent/guardian to understand and comply with the requirements of the protocol and able to fill an appropriate written informed consent.
3. Children and parents who agree to wait for the stipulated time before and after the extraction.

Exclusion Criteria:

1. Children with acute pain.
2. Patients taking analgesics within 5 hours prior to the dental extraction.
3. Patients with a history of prolonged bleeding, platelet disorders, hypersensitivity, or allergic reactions to analgesics or any of the drugs tested.
4. Patients without a home telephone or without parental supervision for the post- operative period.

Ages: 7 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 52 (Estimated)
Dates: Start 2017-05-01 (Actual); Primary Completion 2017-09-01 (Estimated); Study Completion 2017-12-01 (Estimated)

PRIMARY OUTCOMES:
categorical score | 1 hour
  mild, moderate, sever, very sever

SECONDARY OUTCOMES:
binary | 1 day
  yes or no

CONTACTS AND LOCATIONS:
Overall Officials: fatma A. Elshehaby, Professor, Study Director — Cairo University
Locations (1):
- Faculty of Dentistry, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No
i will be available after finished

REFERENCES:
- [Result] Gazal G, Mackie IC. A comparison of paracetamol, ibuprofen or their combination for pain relief following extractions in children under general anaesthesia: a randomized controlled trial. Int J Paediatr Dent. 2007 May;17(3):169-77. doi: 10.1111/j.1365-263X.2006.00806.x. PMID 17397460
- See also: Description paper — https://www.ncbi.nlm.nih.gov/pubmed/21470320